CLINICAL TRIAL: NCT06738758
Title: Multicenter Real-World Cohort Study Evaluating the Impact of Early Intensive Lipid-Lowering Therapy on the Prognosis of Acute Coronary Syndrome Patients
Brief Title: Multicenter Real-World Cohort Study Evaluating the Impact of Early Intensive Lipid-Lowering Therapy on the Prognosis of Acute Coronary Syndrome Patients(ELITE-ACS)
Acronym: ELITE-ACS
Status: Recruiting | Type: Observational
Sponsor: Yun Dai Chen (Other)
Responsible Party: Sponsor-Investigator, Yun Dai Chen, professor, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Other Study IDs: ELITE-ACS
Record Dates: First submitted 2024-12-02; First posted 2024-12-18 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-02

CONDITIONS: Acute Coronary Syndromes
Keywords: Acute Coronary Syndromes; PCSK9 Inhibitor; Lipid compliance time and rate; First cardiovascular event
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Intensive treatment group: patients were treated with PCSK9 inhibitors (with or without statins ± Ezetimibe/Hybutimibe)
  Interventions: Drug: PCSK9 inhibitor
- Conventional combination therapy group: patients were treated with statin＋Ezetimibe/Hybutimibe
  Interventions: Drug: Statin+Ezetimibe/Hybutimibe compound
- control group: patients were treated with statin only
  Interventions: Drug: Statin

INTERVENTIONS:
Drug: PCSK9 inhibitor — The patient used PCSK9 inhibitor (with or without statins ± Ezetimibe/Hybutimibe) in the early hospitalization, and patients continually prescribed or stopped PCSK9 inhibitors treatment during the follow-up visit, which depend on physician's clinical decision and patient preference. PCSK9 inhibitors include Evolocumab, Alirocumab, Tafolecimab, Recaticimab, and Inclisiran, among others.
  Groups: Intensive treatment group
Drug: Statin+Ezetimibe/Hybutimibe compound — The patient used statins and Ezetimibe/Hybutimibe in early hospitalization, and then once a day for 12 months. Whether to adjust the lipid-lowering regimen during follow-up depends on physician's clinical decision and patient preference.
  Groups: Conventional combination therapy group
Drug: Statin — The patient used statins in early hospitalization, and then once a day for 12 months. Whether to adjust the lipid-lowering regimen during follow-up depends on physician's clinical decision and patient preference.
  Groups: control group

SUMMARY:
The purpose of this clinical trial is to evaluate the impact of early initiation of PCSK9 inhibitor therapy for intensive lipid-lowering in Chinese patients with acute coronary syndrome (ACS) during hospitalization on the rate of lipid goal attainment, the time to achieve guideline-recommended lipid levels within one year, and the incidence of adverse cardiovascular events.

The primary research question is whether early initiation of PCSK9 inhibitor therapy during hospitalization for ACS patients in a real-world Chinese setting can increase the rate of lipid goal attainment, shorten the time to reach guideline-recommended lipid levels within one year, and improve the risk of adverse cardiovascular events.

Researchers will compare three lipid-lowering strategies: PCSK9 inhibitor therapy (with or without statins ± Ezetimibe/Hybutimibe), statin plus Ezetimibe/Hybutimibe therapy, and statin monotherapy, to assess the potential of PCSK9 inhibitor drugs in accelerating lipid goal achievement and reducing adverse cardiovascular events in ACS patients.

Participants will:

Receive PCSK9 inhibitor therapy (with or without daily statins ± Ezetimibe/Hybutimibe) every two weeks, or daily statin plus Ezetimibe/Hybutimibe therapy, or daily statin monotherapy.

Undergo follow-up assessments of relevant laboratory indicators at baseline, 3 days after admission, discharge, and 1, 3, 6, and 12 months post-discharge.

Record the occurrence of major adverse cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. This hospitalization for ACS, which includes ST-segment elevation MI (STEMI), non-ST-segment elevation MI (NSTEMI), or unstable angina pectoris (UA) with a GRACE score of intermediate to high risk.
3. Written informed consent must be obtained from eligible patients prior to study enrollment.
4. LDL-C ≥1.8 mmol/L in patients using statin; LDL-C ≥2.6 mmol/L in those not taking statin in the last 4 weeks.

Exclusion Criteria:

1. Received PCSK9 inhibitor therapy within 3 months.
2. Patient has any life-threatening severe disease, including severe liver injury and persistent elevation of serum transaminases, and severe renal failure.
3. Patient has a history of renal or cardiac transplantation.
4. The patient is a pregnant or breastfeeding woman or a woman planning to become pregnant.

Patients judged by the investigator to be unsuitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized for acute coronary syndrome (ACS). ACS is defined as STEMI, NSTEMI, and UA, where UA must be classified as high-risk in the GRACE score.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Lipid attainment rate at each visit node during the observation period (<1.4 mmol/L) | 3 days of medication; At hospital discharge, which is expected to occur between 5 to 10days after admission, depending on the patient's clinical progress; At 1, 3, 6, 12 months after discharge
  Lipid attainment rate at each visit node during the observation period (<1.4 mmol/L)

SECONDARY OUTCOMES:
The average time for different treatment groups to reach the guideline-recommended lipid standards (<1.4mmol/L) during the observation period. | 3 days of medication; At hospital discharge, which is expected to occur between 5 to 10days after admission, depending on the patient's clinical progress; At 1, 3, 6, 12 months after discharge
  The average time for different treatment groups to reach the guideline-recommended lipid standards (<1.4mmol/L) during the observation period.
The overall incidence of the first major adverse cardiovascular events (MACEs) within 12 months in different treatment groups | 12 months
  Description: MACEs was defined as the composite of myocardial infarction, ischemic stroke, cardiovascular death and coronary revascularization
Time from in-hospital initiation of lipid-lowering therapy to first occurrence of any of the above clinical events | 12 months
Percentage change from baseline in LDL-C across treatment groups at different visit nodes | 3 days of medication; At hospital discharge, which is expected to occur between 5 to 10days after admission, depending on the patient's clinical progress; At 1, 3, 6, 12 months after discharge
Change from baseline in inflammatory factors | 3 days of medication; At hospital discharge, which is expected to occur between 5 to 10days after admission, depending on the patient's clinical progress; At 1, 3, 6, 12 months after discharge
  Inflammatory factors include IL-6, CRP/Hypersensitive CRP

OTHER OUTCOMES:
The correlation between LDL-C in-hospital compliance, 1-month compliance, and 3-month compliance with MACE | At hospital discharge, which is expected to occur between 5 to 10days after admission, depending on the patient's clinical progress; At 1, 3, 6, 12 months after discharge
The correlation between the duration of LDL-C within the target and MACE | 12 months
The correlation between different baseline GRACE score levels (low, medium, high) and MACE | 12 months
The correlation between different baseline inflammatory cytokine level groups (quartiles) and MACE | 12 months
The correlation between different baseline age groups (≤ 45 years old or not) and MACE | 12 months
Percentage change in FAI measured by cardiac CT in patients undergoing elective PCI | 12 months
  FAI is a quantitative indicator of inflammation in perivascular adipose tissue measured by CCTA.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China